CLINICAL TRIAL: NCT06238570
Title: Validation of Semi-automatic Oocyte Vitrification by the GAVI® Machine in Medically Assisted Reproduction With Oocyte Donation
Brief Title: Validation of Donor Oocytes Semi-automated Vitrification
Acronym: GAVIDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AOI 2020 CHAPUT
Record Dates: First submitted 2023-02-16; First posted 2024-02-02 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-06

CONDITIONS: Vitrification; Egg Donor; Fertility; Assisted Reproductive Technology
Keywords: Fertility; Egg donor; Vitrification; Assisted Reproductive Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual vitrification (using Vitrolife system) (Placebo Comparator): The vitrification of the oocytes will be carried out by an authorized technician according to the manual protocol validated and used routinely.
  Interventions: Device: Vitrolife system
- Semi-automatic vitrification of oocytes using the GAVI® automaton (Merck) (Active Comparator): The vitrification of the oocytes will be carried out using the GAVI® automaton
  Interventions: Device: Gavi, Merck® (automated vitrification instrument)

INTERVENTIONS:
Device: Gavi, Merck® (automated vitrification instrument) — This instrument recently appeared on the market and demonstrated a high effectiveness in terms of processing time and reproducibility for embryo vitrification. To date, no study has analyzed the efficiency of this automated vitrification instrument on oocyte vitrification.
  The oocytes will be stored in closed cassettes in liquid nitrogen
  Arms: Semi-automatic vitrification of oocytes using the GAVI® automaton (Merck)
Device: Vitrolife system — The oocytes vitrification will be carried out by an authorized technician according to the manual protocol validated and used routinely.
  Arms: Manual vitrification (using Vitrolife system)

SUMMARY:
Oocyte vitrification is an effective method of freezing which has been authorized in France since 2011. The arrival of this technique has led to real improvements in the survival rate of oocytes after warming compared to that observed after slow freezing, a method previously applied. Oocytes reheated after vitrification show excellent results in terms of vitality and recovery of cellular functionality. Indeed, the fertilization rates observed after using warmed and fertilized oocytes in Assisted Reproduction Technology (ART) by intracytoplasmic sperm injection (ICSI) are similar to those obtained with fresh oocytes.

However, the manual vitrification techniques used until now involve a learning curve and a potential variability of the completion time depending on the operator and the number of oocytes to be vitrified.

Oocyte vitrification is a key step to optimize the chances of pregnancy in ART after using these oocytes. However, manual vitrification requires a learning curve, is technician-dependent and requires significant technical time.

A semi-automatic vitrification device (GAVI®, Merck), which recently appeared on the market, has demonstrated its effectiveness in terms of speed of production and reproducibility of vitrification of embryos obtained in ART. To our knowledge, no study has analyzed the effectiveness of semi-automatic vitrification (GAVI®, Merck) on survival and oocyte quality after warming. It would therefore be interesting to evaluate the effectiveness of this automaton on oocyte vitrification in the context of oocyte donation and to determine the impact of semi-automatic vitrification on oocytes compared to manual vitrification.

The main objective of this study is to demonstrate the non-inferiority of vitrification semi-automated device (Gavi) of oocytes with regard to the oocyte survival rate, compared to the manual technique used in ART.

The investigator will compare the effectiveness of semi-automated vitrification device with the manual technique, in terms of ART results by comparing the fertilization rates, the number and quality of embryos obtained as well as the implantation rates in oocyte recipient patients. This study will then allow clinical application of the most efficient protocol for oocyte vitrification in the context of oocyte donation. A cost/effectiveness study will be carried out.

DETAILED DESCRIPTION:
The oocytes will be stored in closed devices (Rapid I® straws for the manual vitrification protocol or pods® in cassettes for the semi-automatic vitrification protocol) in liquid nitrogen. All samples are anonymized in the context of oocyte donation by the medically assisted procreation (PMA) department of Clermont-Ferrand University Hospital, according to the method usually used.

The oocyte survival rate will be evaluated by the service technician or biologist. This survival rate corresponds to the ratio between the number of oocytes intact 2 hours after warming and able to be microinjected with a spermatozoon (ICSI), and the number of oocytes heated, after vitrification. We will compare the oocyte survival rate after vitrification and semi-automatic warming vs. after manual vitrification.

The investigator will compare the effectiveness of ART with oocyte donation during semi-automatic vitrification of oocytes compared to the manual technique, with regard to:

* Oocyte functional quality after warming evaluated by the fertilization rate of oocytes after ICSI
* Early development of embryos:

  * the number of embryos cleaved on the 2nd day of culture from vitrified oocytes, the blastulation rate defined by the ratio between the number of blastocysts obtained (Gardner classification on the 5th day of culture) and the total number of cleaved embryos.

These parameters will be assessed daily during the embryo reading by a technician or a biologist from the ART department.

We will also compare the effectiveness of ART with oocyte donation during the semi-automatic vitrification of oocytes compared to the manual technique, with regard to:

* The implantation rate of embryos from vitrified oocytes, defined by the ratio between the number of embryo sacs observed (6th week of amenorrhea) and the number of embryos transferred
* The rate of miscarriages in oocyte recipients. These parameters will be evaluated by a biologist from the ART department after the results of the beta hCG of the patients and the performance of the ultrasound at the 6th week of amenorrhea by the gynecologists of the ART department.

ELIGIBILITY:
Inclusion Criteria:

* Egg donor
* Oocyte puncture for donation
* Good quality ovarian reserve (Antral follicle count evaluated by ultrasound: CFA ≥ 7)
* Negative serology status (HIV, hepatitis B and C, syphilis, CMV and HTLV)
* Absence of symptoms or COVID contact
* Absence of genetic contraindication to egg donation
* Woman able to give informed consent to participate in research
* Woman affiliated to a social security scheme

Exclusion Criteria:

* Decline to participate
* Pregnant and lactating woman
* Person under guardianship, curatorship, deprivation of liberty, protection of justice

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Oocyte survival | two years after the inclusion
  Oocyte survival after semi-automated vitrification by the GAVI® device compared to the manual technique (Vitrolife) with egg donation. A warmed oocyte that has survived can then be used in AMP by ICSI technique.

SECONDARY OUTCOMES:
Effectiveness of ART with egg donation after oovcytes semi-automated vitrification | two years after vitrification
  * oocyte functional quality after warming by assessing the fertilization rate for each oocyte
  * early development of embryos: number of embryos cleaved on the 2nd day of culture from vitrified oocytes, blastulation rate defined by the ratio between the number of blastocysts obtained (Gardner classification on the 5th day of culture) and total number of cleaved embryos.
  * implantation rate of embryos from vitrified oocytes, defined by the ratio between the number of embryonic sacs observed (6th week of amenorrhea) and the number of embryos transferred
  * rate of miscarriages in egg recipients
Study the costs and cost-effectiveness | at the end of the study 24 months
  Study the costs and cost-effectiveness of ART by egg donation, during semi-automatic oocyte vitrification and during manual technique, from a hospital point of view.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France